CLINICAL TRIAL: NCT02058836
Title: Botulinum Toxin for the Management of Chronic Orchialgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00023188
Record Dates: First submitted 2014-02-05; First posted 2014-02-10 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Chronic Testicular Pain
Keywords: Chronic testicular pain; Orchialgia; Botulinum toxin; Botox; Urology
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Botox Injection (Experimental): The participant will be given an injection of Botox along the spermatic cord under ultrasound guidance. Before drug administration, a nerve block using bupivacaine will be completed to numb the area for treatment. This will be a 10 mL injection done one time at the initial patient visit.
  Interventions: Drug: Botox Injection
- Saline Injection (Placebo Comparator): The patient will receive an inactive injection of normal saline along the spermatic cord under ultrasound guidance. This will be a 10 ml injection done once at the initial visit. Before the injection of saline, a spermatic cord block using bupivacaine will be completed to numb the area for treatment.
  Interventions: Procedure: Normal saline injection

INTERVENTIONS:
Drug: Botox Injection — One-time injection of 100 Units of Botox in 10 mL of saline. The 10 mL injection will be distributed in 4 areas around the spermatic cord and testicle of the affected side with 2.5 mL being injected at each area.
  Other Names: Botox; Botulinum toxin-A
  Arms: Botox Injection
Procedure: Normal saline injection — One-time injection of 10 mL of 0.9% sodium chloride (normal saline) solution. The 10 mL injection will be distributed in 4 areas around the spermatic cord and testicle of the affected side with 2.5 mL being injected at each area.
  Other Names: 0.9% Sodium Chloride injection; Saline injection
  Arms: Saline Injection

SUMMARY:
The purpose of this research study is to determine if Botox injections will provide relief from chronic testicular pain. In the study, the spermatic cord of particpants will be injected with either Botox or a placebo of saline. Botox is currently used to treat other urological conditions like overactive bladder and lower urinary tract problems. For these conditions, Botox works by relaxing muscles in the affected areas. The investigators believe that Botox will act similarly in the treatment chronic testicular pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic testicular pain (orchialgia)

Exclusion Criteria:

* Active infection of urinary tract (UTI)
* Active infection of the scrotal skin of the affected side
* Bilateral orchiectomy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10-18 (Actual); Study Completion 2016-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Terlecki, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botox Injection | Saline Injection
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox Injection | Saline Injection | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.25 (8.14) | 56.25 (12.5) | 65.75 (14.10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale for Pain Score
Description: Visual Analog Scale for Pain Score (VAS). It measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms such as pain. VAS is a straight horizontal line of fixed length, usually 100 mm. The patient marks on the line the point that they feel represents their perception of their current state.The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks. The score range is from 0-100. Lower scores denotes better outcomes.
Time Frame: Baseline and 1 Week Post Injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units on a scale
  Baseline | 59.3 (17.6) | 30.3 (16.4)
  1 Week Post Procedure | 55.0 (22.9) | 75.0 (7.8)

2. Primary Outcome: Visual Analog Scale for Pain Score
Description: Visual Analog Scale for Pain Score. It measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms such as pain. VAS is a straight horizontal line of fixed length, usually 100 mm. The patient marks on the line the point that they feel represents their perception of their current state.The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks. The score range is from 0-100. Lower scores denotes better outcomes.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units on a scale
  Baseline | 59.3 (17.6) | 30.3 (16.4)
  1 Month Post Procedure | 56 (31.5) | 72.7 (30.0)

3. Primary Outcome: Visual Analog Scale for Pain Score
Description: as for outcome 2
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units on a scale
  Baseline | 59.3 (17.6) | 30.3 (16.4)
  3 Months Post Procedure | 63 (20.6) | 84 (3.5)

4. Primary Outcome: Visual Analog Scale for Pain Score
Description: as for outcome 2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units on a scale
  Baseline | 59.3 (17.6) | 30.3 (16.4)
  6 Months Post Procedure | 78.7 (12.1) | 61 (29.5)

5. Primary Outcome: Quality of Life Questionnaire Score
Description: Quality of Life Questionnaire Score (QOL). To assess the QOL, a short form-36 (SF-36) was used. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. The SF-36 consists of eight items, which are the weighted sums of the questions in their section. The eight items are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. Items in the same scale are averaged together to create the 8 scale scores. Scale scores represent the average for all items in the scale that the respondent answered. Higher scores denotes better outcomes.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 2
units on a scale | 67.41 (18.27) | 84.31 (6.48)

6. Primary Outcome: Quality of Life Questionnaire Score
Description: Quality of Life Questionnaire Score. To assess the QOL, a SF-36 was used. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The score range is 0-100 and higher scores denotes better outcomes.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units on a scale | 66.48 (33.40) | 83.66 (14.94)

7. Primary Outcome: Quality of Life Questionnaire Score
Description: as for outcome 5
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units on a scale | 67.56 (30.90) | 84.44 (11.46)

8. Primary Outcome: Quality of Life Questionnaire Score
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units on a scale | 77.04 (14.29) | 86.59 (9.23)

9. Primary Outcome: Units of Analgesics Used for Testicular Pain
Description: Change from Baseline in Units of Analgesics Used for Testicular Pain
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units of analgesics
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units of analgesics
  Baseline | 3.3 (5.77) | 2.5 (2.5)
  1 Week Post Procedure | 1.7 (2.9) | 2.1 (2.6)

10. Primary Outcome: Units of Analgesics Used for Testicular Pain
Description: Change from Baseline in Units of Analgesics Used for Testicular Pain
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units of analgesics
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units of analgesics
  Baseline | 3.3 (5.77) | 2.5 (2.5)
  1 Month Post Procedure | .13 (.23) | 2.1 (2.6)

11. Primary Outcome: Units of Analgesics Used for Testicular Pain
Description: Change from Baseline in Units of Analgesics Used for Testicular Pain
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units of analgesics
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units of analgesics
  Baseline | 3.3 (5.77) | 2.5 (2.5)
  3 Months Post Procedure | .67 (1.2) | 2 (2.6)

12. Primary Outcome: Units of Analgesics Used for Testicular Pain
Description: Change from Baseline in Units of Analgesics Used for Testicular Pain
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units of analgesics
Arm/Group | Botox Injection | Saline Injection
Number analyzed (Participants) | 3 | 3
units of analgesics
  Baseline | 3.3 (5.77) | 2.5 (2.5)
  6 Months Post Procedure | 0 (0) | 2.5 (2.5)

ADVERSE EVENTS:
Arm/Group | Botox Injection | Saline Injection
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes